CLINICAL TRIAL: NCT04126551
Title: Unraveling the Role of Mitochondrial DNA Methylation in Type 2 Diabetes
Brief Title: Mitochondrial Methylation in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Dawn K Coletta, Associate Professor of Medicine, University of Arizona
Other Study IDs: 1901254125
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Overweight; Obesity; Diabetes Mellitus, Type 2; Insulin Resistance
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from vastus lateralis skeletal muscle biopsies and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lean, healthy control: Lean, healthy control subjects. Volunteers will be matched for sex and age 21-55 years old. Ethnicities studied will be self-reported. We will attempt to match on race/ethnicities with equal numbers of non-Hispanic/Latinos and Hispanics/Latinos.
  Interventions: Other: Methylation status
- Overweight/obese nondiabetic: Overweight/Obese nondiabetic subjects. Overweight and obesity will be defined using the standard body mass index cutoffs. Volunteers will be matched for sex and age 21-55 years old. Ethnicities studied will be self-reported. We will attempt to match on race/ethnicities with equal numbers of non-Hispanic/Latinos and Hispanics/Latinos.
  Interventions: Other: Methylation status
- Type 2 diabetes: Participants with type 2 diabetes will be diagnosed accordingly to ADA criteria. Volunteers will be matched for sex and age 21-55 years old. Ethnicities studied will be self-reported. We will attempt to match on race/ethnicities with equal numbers of non-Hispanic/Latinos and Hispanics/Latinos.
  Interventions: Other: Methylation status

INTERVENTIONS:
Other: Methylation status — Participants will be recruited, and muscle biopsies will be obtained for methylation analyses and measuring mitochondrial function

SUMMARY:
The overarching goal of this proposal is to determine whether DNA methylation of the mitochondrial DNA impairs mitochondrial function in insulin resistant states such as overweight/obesity and type 2 diabetes.

DETAILED DESCRIPTION:
To determine whether differences in human skeletal muscle DNA methylation patterns in the mitochondrial and nuclear genome can explain the lower abundance of ETC and OXPHOS mRNA and protein observed in insulin resistant skeletal muscle of overweight/obese and type 2 diabetic participants. To determine whether patterns of human skeletal muscle DNA methylation in the mitochondrial and nuclear genome are predictive of ETC function. We will isolate skeletal muscle mitochondria from metabolically well-characterized lean insulin sensitive, overweight/obese insulin resistant nondiabetic and obese insulin resistant type 2 diabetic volunteers, and functionally evaluate each ETC complex (I - IV) and complex V (ATP synthase).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 21-55 years old
2. Body Mass Index:

   Lean, healthy BMI ≤25; Overweight,non-diabetic BMI 25-29.9; Obese, non-diabetic BMI 30-50; Type 2 Diabetes (per the American Diabetes Association criteria)
3. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
4. Female subjects must be non-lactating and will be eligible only if they have a negative pregnancy test throughout the study period, and must agree to use acceptable birth control (hormonal contraceptives, barrier methods, have an intrauterine device, or surgical sterilization)
5. Subjects must have the following laboratory values:

   * Hematocrit ≥ 35 vol%
   * Serum creatinine ≤ 1.6 mg/dl
   * AST (SGOT) < 2 times upper limit of normal
   * ALT (SGPT) < 2 times upper limit of normal
   * Alkaline phosphatase < 2 times upper limit of normal
   * Triglycerides < 150 mg/dl for nondiabetics
   * Triglycerides <300 for diabetics
   * INR ≤ 1.3
   * HbA1c ≤ 10

Exclusion Criteria:

1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on a stable dose of such agents for the past three months before entry into the study. Subjects must not be taking estrogens or other hormonal replacement therapy unless the subject has been on these agents on a stable dose for the prior three months. Subjects taking systemic glucocorticoids are excluded. Patients with type 2 diabetes will be excluded if they are taking thiazolidinediones.
2. Subjects receiving Gemfibrozil must not also be receiving a statin.
3. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
4. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP>160, diastolic BP>95, autonomic neuropathy, resting heart rate >100, electrolyte abnormalities.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups of volunteers will be studied: 1) lean, healthy volunteers, 2) overweight/obese volunteers without type 2 diabetes, and 3) volunteers with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mitochondrial DNA methylation | 3 years
  Mitochondrial DNA methylation and D-loop of mitochondria is altered in insulin resistant states such as overweight/obesity and type 2 diabetes

SECONDARY OUTCOMES:
Mitochondrial Function | 3 years
  The extent of mitochondrial function impairment in insulin resistant participants corresponds to the degree of methylation of the mitochondrial genome and D-loop

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Coletta, PhD, Principal Investigator — University of Arizona
Locations (1):
- Clinical and Translational Research Center (CaTS), Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No